CLINICAL TRIAL: NCT07348276
Title: First-in-Human Study for the Safety and Evaluation of Two 4R Tau Ligands ([18F]ABBV964i and [ 18F]ABBV-965i) as Potential PET Radioligands for Imaging Tau Protein in the Brain of Patients With Probable PSP and Healthy Volunteers
Brief Title: First-in-Human Study for the Safety and Evaluation of Two 4R Tau Ligands as Potential PET Radioligands for Imaging Tau Protein in the Brain
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Collaborators: Enigma Biomedical USA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: EPAA-2024-TR01
Record Dates: First submitted 2025-12-26; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Progressive Supranuclear Palsy (PSP); Healthy Participants
Keywords: Tauopathy; Tau; PET Imaging; ABBV-965i; ABBV-964i; PSP; Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Tauopathies; Pick Disease of the Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Dosimetry (Experimental): Healthy participants receive [18F]ABBV-964i and [18F]ABBV-965i for PET imaging.
  Interventions: Drug: [18F]ABBV-964i; Drug: [18F]ABBV-965i
- Part B - Proof of Concept (Experimental): Participants receive [18F]ABBV-964i and [18F]ABBV-965i for PET imaging to see how the drugs work in the brain.
  Interventions: Drug: [18F]ABBV-964i; Drug: [18F]ABBV-965i
- Part C - Test-Retest (Optional) (Experimental): Participants receive two PET scans using the same drug to see if results are consistent.
  Interventions: Drug: Lead Candidate

INTERVENTIONS:
Drug: [18F]ABBV-964i — PET radiopharmaceuticals selective for tau, administered intravenously at doses up to 10 mCi.
  Arms: Part A - Dosimetry; Part B - Proof of Concept
Drug: [18F]ABBV-965i — PET radiopharmaceuticals selective for tau, administered intravenously at doses up to 10 mCi.
  Arms: Part A - Dosimetry; Part B - Proof of Concept
Drug: Lead Candidate — Preferred PET radiopharmaceuticals (between [18F]ABBV-964i and [18F]ABBV-965i) selective for tau, administered intravenously at doses up to 10 mCi.
  Other Names: [18F]ABBV-965i; [18F]ABBV-964i
  Arms: Part C - Test-Retest (Optional)

SUMMARY:
This clinical study is being conducted to learn more about two new imaging drugs, called [18F]ABBV-964i and [18F]ABBV-965i, which are designed to help doctors see changes in the brain related to a condition called Progressive Supranuclear Palsy (PSP). PSP is a rare disease that affects movement, balance, and thinking. These drugs are used with a type of scan called PET (Positron Emission Tomography) to show areas of the brain where a protein called tau builds up. Tau buildup is linked to PSP and other brain diseases.

The main goal of this study is to find out if these imaging drugs are safe for people and if they work well to show tau in the brain. The study will also look at how the drugs move through the body and how much radiation they give off. Researchers hope this information will help develop better tools for diagnosing PSP and tracking how it changes over time.

Who can join? Adults who are healthy or who have PSP may be able to take part. Participants will have screening tests to make sure they qualify.

What does participation involve? People in the study will have PET scans, blood tests, and other safety checks. Some participants will also have an MRI scan. The study is divided into three parts: Part A checks radiation levels in healthy volunteers, Part B looks at how the drugs work in the brain of PSP patients and healthy volunteers, and Part C (optional) repeats scans to see if results are consistent.

Why is this important? There is currently no cure for PSP, and better imaging tools could help researchers develop new treatments. By joining this study, participants will help advance research that may improve care for people with PSP and similar conditions in the future.

DETAILED DESCRIPTION:
This Phase 1, first-in-human study is designed to evaluate the safety, pharmacokinetics, biodistribution, and test-retest variability of two investigational PET radioligands, [18F]ABBV-964i and [18F]ABBV-965i, for imaging 4R Tau pathology in individuals with Progressive Supranuclear Palsy (PSP) and healthy volunteers (HV). The study is structured into three parts: Part A (Dosimetry), Part B (Proof-of-Concept), and Part C (Optional Test-Retest).

Part A involves low-dose whole-body PET imaging in HVs to determine radiation dosimetry using both tracers. Participants will receive intravenous injections of [18F]ABBV-964i and [18F]ABBV-965i in separate imaging sessions, followed by dynamic PET acquisitions and urine collection for dosimetry analysis. Dosimetry calculations will employ MIRD methodology and OLINDA software to estimate absorbed organ doses and effective whole-body dose.

Part B evaluates tracer kinetics and brain uptake in PSP and HV participants using dynamic brain PET imaging over approximately 120 minutes post-injection. Arterial and/or venous blood sampling will be performed for kinetic modeling, including radiometabolite analysis via HPLC and plasma free fraction determination. Quantitative modeling will include compartmental approaches and graphical methods, as well as simplified reference tissue models. Key metrics such as SUV, SUVR, VT, and DVR will be derived to characterize tracer binding and distribution. MRI co-registration will support VOI definition for regional analysis.

Part C, if conducted, will assess test-retest reproducibility of the selected tracer in PSP participants using repeated brain PET scans under similar conditions. Variability will be expressed as percentage difference between test and retest values for primary imaging endpoints.

Radiotracer administration will follow strict safety protocols, including dose limits (≤ 10 mCi per injection) and radiation exposure monitoring to ensure compliance with applicable guidelines. PET imaging will be performed on PET/CT systems with attenuation correction. Image reconstruction will utilize OSEM algorithms with scatter and random corrections applied.

Safety assessments include continuous AE monitoring, vital signs, ECGs, and laboratory evaluations at predefined timepoints. Participants will undergo screening procedures including MRI (for PSP), MMSE, PSPRS, and p-Tau217 plasma testing where applicable. Concomitant medications and procedural details (arterial line placement, Allen's test, infusion protocols) are specified to minimize risk and ensure scientific integrity.

The investigational tracers are formulated as sterile solutions for IV injection. Manufacturing and quality control will adhere to GMP standards. The study rationale emphasizes the need for selective 4R Tau imaging agents to advance diagnostic and therapeutic strategies for PSP and related tauopathies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females: PSP 40-80 years; HV 18-80 years
* Body weight: 43-120 kg (95-265 lb)
* Women of childbearing potential: abstinent or use 2 contraception methods (one barrier) during study and 30 days post last injection
* Men: use 2 contraception methods and refrain from sperm donation during study and 90 days post last injection
* Adequate circulation and normal clotting for arterial cannulation
* Sufficient mobility and ability to lie still for imaging
* Healthy Volunteers: informed consent, no clinically relevant findings, no cognitive impairment
* PSP Participants: informed consent or assent with LAR consent, clinical diagnosis per NINDS-SPSP criteria, MRI consistent with PSP, able to ambulate, tolerate MRI, comply with study procedures, caregiver available if needed

Exclusion Criteria:

* History of drug or alcohol abuse in past 12 months
* Clinically significant lab abnormalities or unstable illness
* Investigational drug/device use within 30 days
* Pregnant, lactating, or breastfeeding
* Significant comorbid conditions (GI, CV, hepatic, renal, etc.)
* Abnormal clotting parameters (if arterial sampling)
* MRI contraindications (implants, claustrophobia) for PSP participants
* Use of OTC meds or supplements within 2 weeks (healthy volunteers)
* Use of anti-hemostasis meds within 2 weeks of arterial line placement for PSP participants
* Unable to lie still for 90 minutes
* Major surgery or significant blood loss within 4 weeks
* Positive for Hepatitis B, Hepatitis C, or HIV
* Deemed unsuitable by Investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety of [18F]ABBV-964i and [18F]ABBV-965i: Incidence of Adverse Events | Up to 13 weeks
  Incidence of adverse events (AEs) following administration of [18F]ABBV-964i and [18F]ABBV-965i.
Radiation dosimetry of [18F]ABBV-964i and [18F]ABBV-965i | Up to 13 weeks
  Radiation absorbed dose estimates following administration of [18F]ABBV-964i and [18F]ABBV-965i, derived from PET imaging and dosimetry calculations.

SECONDARY OUTCOMES:
Brain Uptake measured as Standardized Uptake Value (SUV) or equivalent | Up to 13 weeks
  Quantitative assessment of uptake in brain regions measured by PET imaging.
Model-derived Pharmacokinetics parameters | Up to 13 weeks
  Pharmacokinetic parameters of radiotracers derived from dynamic PET imaging and input functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Invicro (dba Perceptive), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided